CLINICAL TRIAL: NCT07189169
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Clinical Study of the Efficacy and Safety of QA108 Granules in the Treatment of Intermediate Age-Related Macular Degeneration (Type of Yang-Hyperactivity Due to Yin-Deficiency)
Brief Title: QA108 Phase III Study in Subjects With Intermediate AMD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Smilebiotek Zhuhai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QA108-III
Record Dates: First submitted 2025-09-14; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Intermediate Age-Related Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QA108 granules, 7.5 g/bag,2 bags/time, BID (Experimental)
  Interventions: Drug: QA108 granules
- QA108 granule simulants, 7.5 g/bag,2 bags/time, BID (Placebo Comparator)
  Interventions: Drug: QA108 granules placebo

INTERVENTIONS:
Drug: QA108 granules — Take the medication as required for 24 weeks
  Arms: QA108 granules, 7.5 g/bag,2 bags/time, BID
Drug: QA108 granules placebo — Take the medication as required for 24 weeks
  Arms: QA108 granule simulants, 7.5 g/bag,2 bags/time, BID

SUMMARY:
This is a phase III randomized, double-masked, placebo-controlled, multicenter study. To evaluate the efficacy and safety of QA108 granules in the treatment of intermediate age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. The study eye meets the Western medicine diagnostic criteria for intermediate age-related macular degeneration;
2. Presence of at least one large drusen (diameter ≥125 μm) in the macular area of the fundus;
3. Consistent with the TCM diagnosis of type of Yang-hyperactivity due to Yin-deficiency;
4. Age 45-85 years (inclusive), regardless of gender;
5. The study eye has a BCVA of 88-34 letters (using the ETDRS chart, inclusive of threshold values), equivalent to a Snellen visual acuity of 20/20 to 20/200 (inclusive);
6. Voluntary participation in this clinical trial, with informed consent provided and an informed consent form signed

Exclusion Criteria:

1. The study eye is with concomitant eye disorders that may interfere with the observation of the trial as judged by the investigator, including pathological myopia, glaucoma, diabetic retinopathy, retinal vein occlusion, uveitis, retinal detachment, optic neuropathy (optic neuritis, atrophy, papilledema), and macular hole;
2. The study eye has an intraocular pressure (IOP) ≥ 25 mmHg;
3. Presence of geographic atrophy (GA) involving the foveal center in the study eye;
4. Previous ophthalmic surgery in the study eye: vitrectomy, macular translocation;
5. Aphakia (except pseudophakia) or posterior capsule rupture (except YAG laser posterior capsulotomy after IOL implantation at more than 1 month prior to screening) of the study eye;
6. Any intraocular surgery (excluding intravitreal injections) that may affect trial observations or imaging in the study eye within 3 months;
7. Cataract in the study eye that interferes with fundus examination or imaging;
8. Treatments received in the study eye within 3 months prior to screening, including macular laser photocoagulation and micropulse laser therapy;
9. The patient received relevant TCM treatment within 1 month prior to screening;
10. Active ocular infection in either eye that affects fundus examination or imaging;
11. The non-study eye has a BCVA of less than 19 ETDRS letters (not inclusive);
12. Known allergy to the therapeutic or diagnostic drug used in the study protocol, including the single drug components in the study drugs;
13. Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg after regular use of antihypertensive drugs);
14. Platelet count ≤100×10⁹/L (unless follow-up results are normal), or any of the following exceeding 1.5 times the upper limit of normal (ULN): total bilirubin (TBIL), alanine aminotransferase (ALT), aspartate aminotransferase (AST), or serum creatinine (Cr);
15. Pregnant women, women who are breastfeeding, those who plan for pregnancy in the next six months, or those who are unwilling to take effective birth controls during the study course and until six months after drug withdrawal;
16. Any uncontrollable clinical disorder prior to the start of treatment, such as severe psychiatric, neurological, respiratory, immunological, hematological, and cardiac system diseases, and malignant tumors;
17. Subjects who have participated in other clinical trials within 3 months prior to this trial;
18. Patients who are unsuitable for participating at the discretion of the investigator.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in drusen area | weeks 24

SECONDARY OUTCOMES:
Percentage change from baseline in drusen area | weeks 12

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, China